CLINICAL TRIAL: NCT04763135
Title: What is the Effectiveness and Safety of Mirtazapine Versus Escitalopram in Alleviating Cancer-associated Poly-symptomatology (MIR-P)? A Mixed-method Randomized Controlled Trial Protocol
Brief Title: Mirtazapine in Cancer-related Poly-symptomatology
Acronym: MIR-P
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: difficulties in recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL20_0032; 2020-002994-90 (EudraCT Number)
Record Dates: First submitted 2021-02-15; First posted 2021-02-21 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Cancer; Neoplasms; Neoplasm Metastasis
Keywords: Cancer; Symptom management; Poly-Symptomatology; Mirtazapine; Antidepressive drugs
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — Mirtazapine; Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral mirtazapine (Experimental): Arm 1 patients will be treated using a daily mirtazapine treatment. Treatment will be taken on the evening. Treatment will be initiated at 15 mg daily and gradually increased depending on symptom control and side effects. Treatment doses will be adapted for old patients and those with liver failure.
  Interventions: Drug: Mirtazapine
- Oral escitalopram (Active Comparator): Arm 2 patients will be treated using a daily escitalopram treatment. Treatment will be taken in the morning. Treatment will be initiated at 10 mg daily and gradually increased depending on symptom control and side effects. Treatment doses will be adapted for 5 mg for old patients.
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Mirtazapine — Orally disintegrating tablets of mirtazapine introduced at the dose of 15 mg and increased up to 45 mg per day during 56 days.
  Doses escalation: based on symptom management and side effect assessment.
  Arms: Oral mirtazapine
Drug: Escitalopram — Orally disintegrating tablets of escitalopram introduced at the dose of 10 mg (or 5 mg for patients older than 65) and increased up to 20 mg per day during 56 days.
  Doses escalation: based on symptom management and side effect assessment.
  Arms: Oral escitalopram

SUMMARY:
Multicenter, prospective, randomized, controlled trial based on a mixed-method methodology using parallel groups, of oral mirtazapine (intervention) compared with oral escitalopram (control), with a 56 days follow-up. Improvement of the Global health Status (issued from the EORTC-QLQ-C30 (Quality of Life Questionnaire)) will be used as the primary outcome on day 56. Semi-structures interviews will be performed on a purposive sample for qualitative analysis. The 418 participants will be followed-up at day 7, 14, 28 and 56 for a 56 days period. A sub-group of participants will be invited to take part into qualitative interviews at baseline and day 56. Recruitment of participants to the qualitative part will be based on a purposive sampling.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* Suffering from advanced cancer
* Having a clinically estimated life expectancy over 3 months.
* Being diagnosed from having a depressive syndrome by a Hospital Anxiety and Depression Scale-D over 11.
* Being in need of an antidepressant treatment.
* Suffering from at least one under-controlled symptom (defined as a score over 3 on the Edmonton Symptom Assessment Scale) among: pain, nausea, vomiting, breathlessness, lack of appetite, sleep disorders, anxiety or impaired wellbeing.
* Having or not a cancer treatment.
* Being able to understand the information related to the study, and to sign informed consent.
* Having agreed to take part to the study.
* Being able to fill Patient Reported Outcomes questionnaires.
* Being available to be call on days 7 and 14.
* Having a social security affiliation.

Exclusion Criteria:

* Being treated by an antidepressive agent during the four weeks before inclusion.
* Having had a hypersensitivity event to mirtazapine, escitalopram of any excipient.
* Having had a prior inefficient treatment by mirtazapine or escitalopram.
* Having postural hypotension or arterial systolic hypotension inferior to 90 mmHg measured following the guidelines of the European Society of Cardiology
* Having a QT interval over 420 ms.
* Having uncontrolled hearth rhythm disorder or uncontrolled conduction disorder.
* Having had or having bipolar disorder.
* Having uncontrolled seizure or epilepsy (relative non-inclusion criteria needing a neurology specialist opinion)
* Having or having history of closed-angle glaucoma.
* Having bone marrow aplasia.
* Practicing breast-feeding or being pregnant.
* Women of childbearing age with no contraception method.
* Having a treatment with:
* Monoamine oxidase inhibitors (Selegiline, Moclobemide, Isocarboxazid, Nialamide, Phenelzine, Tranylcypromine, Iproniazid, Iproclozide, Toloxatone, Linezolid, Safinamide, Rasagiline)
* One of the following antiarrhythmic drugs: Flecainide, Propafenone, any class IA and III antiarrhythmic drug (amiodarone, disopyramide, hydroquinidine, quinidine, procainamide, sparteine, ajmaline, prajmaline, lorajmine, bretylium tosilate, bunaftine, dofetilide, ibutilide, tedisamil, dronedarone).
* Linezolid, sparfloxacin, moxifloxacin, macrolides (IV erythromycin, josamycin, clarithromycin, telithromycin), pentamidin, halofantrine, HIV protease inhibitors (ritonavir, nelfinavir, amprenavir, indinavir), azolic antifungal agents (ketoconazole, itraconazole, miconazole, fluconazole, voriconazole)
* Mizolastine and Astémizole
* St. John's wort
* Having genetic galactose intolerance or glucose-galactose malabsorption.
* Having one of the following electrolyte disorders not corrected at the time of inclusion: hyponatremia, hyperkalemia, hypokalemia, hypermagnesemia, and hypomagnesemia.
* Having end-stage renal disease with a creatinine clearance inferior to 15 ml/min calculated using the Cockroft's formula.
* Having hepatic failure.
* Having legal incapacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
Global health status score | At baseline and day 56
  The Global Health Status will be calculated from the specific subscale included in the EORTC-QLQ-C30 scale.
  The difference between baseline and the end-point (day 56) will be the primary judgment criteria. A 4 to 8 points difference between baseline and endpoint will be considered as a mild difference, and a difference over 8 points will be considered as a moderate difference.

SECONDARY OUTCOMES:
The subjective experience associated with symptoms burden. | At baseline and day 56.
  Qualitative analysis of compared semi-structured interviews undertaken at baseline and day 56 on a convenience sample.
Proportion of mitigated symptoms. | Day 28
  The Edmonton Symptom Assessment Scale 12F will be used to assess each symptoms intensities for the following symptoms: pain, nausea, vomiting, lack of appetite, breathlessness, depression, anxiety, sleep disorders and wellness.
  For each symptom, the difference between baseline and the assessment time will be calculated. A difference equal or over one point will be regarded as mitigation. The judgment criteria will be the proportion of symptoms that were rated over three at baseline and that were mitigated at the assessment time.
Proportion of mitigated symptoms. | Day 56
  The Edmonton Symptom Assessment Scale 12F will be used to assess each symptoms intensities for the following symptoms: pain, nausea, vomiting, lack of appetite, breathlessness, depression, anxiety, sleep disorders and wellness.
  For each symptom, the difference between baseline and the assessment time will be calculated. A difference equal or over one point will be regarded as mitigation. The judgment criteria will be the proportion of symptoms that were rated over three at baseline and that were mitigated at the assessment time.
Auto-assessment depression score. | Day 28
  The Hospital Anxiety and Depression Scale-D auto-assessment score will be used to assess the auto-assessment depression score.
  The judgment criteria will be the difference between baseline and the assessment time. A difference over 1.5 points will be regarded as clinically significant.
Auto-assessment depression score. | Day 56
  The Hospital Anxiety and Depression Scale-D auto-assessment score will be used to assess the auto-assessment depression score.
  The judgment criteria will be the difference between baseline and the assessment time. A difference over 1.5 points will be regarded as clinically significant.
Hetero-assessment-based depression score. | Day 28
  The Montgomery-Asberg Depression Rating Scale hetero-assessment score will be used to assess the hetero-assessment depression score.
  The judgment criteria will be the difference between baseline and the assessment time. A difference over 1.9 points will be regarded as clinically significant.
Hetero-assessment-based depression score. | Day 56
  The Montgomery-Asberg Depression Rating Scale hetero-assessment score will be used to assess the hetero-assessment depression score.
  The judgment criteria will be the difference between baseline and the assessment time. A difference over 1.9 points will be regarded as clinically significant.
Weight control | Day 28
  Weight control will be defined as a difference under 500g between the weight at baseline minus the weight at the assessment time.
  The judgment criteria will be the proportion of patients with weight control at assessment time.
Weight control | Day 56
  Weight control will be defined as a difference under 500g between the weight at baseline minus the weight at the assessment time.
  The judgment criteria will be the proportion of patients with weight control at assessment time.
Weight improvement. | Day 28
  Weight improvement will be defined as a difference over 500g between the weight at the assessment time minus the weight at baseline.
  The judgment criteria will be the proportion of patients with weight improvement at assessment time.
Weight improvement. | Day 56
  Weight improvement will be defined as a difference over 500g between the weight at the assessment time minus the weight at baseline.
  The judgment criteria will be the proportion of patients with weight improvement at assessment time.
Stability in oral morphine milligram equivalents. | Day 28
  The stability in oral morphine milligrams equivalent will be defined as a decrease or stability in the daily doses of opioid pain killers measured using oral morphine milligram equivalents.
  The judgment criteria will be the proportion of patients with stability in oral morphine milligram equivalents.
Stability in oral morphine milligram equivalents. | Day 56
  The stability in oral morphine milligrams equivalent will be defined as a decrease or stability in the daily doses of opioid pain killers measured using oral morphine milligram equivalents.
  The judgment criteria will be the proportion of patients with stability in oral morphine milligram equivalents.
Escalation in symptom control treatment doses | Day 28
  Escalation in symptom control treatment doses will be defined as any escalation in the dose of a treatment existing at baseline or any new treatment introduced to control one of the following symptoms: pain, nausea, vomiting, lack of appetite, breathlessness, depression, anxiety, sleep disorders and wellness.
  The judgment criteria will be the proportion of patients with an escalation in symptom control treatment doses.
Escalation in symptom control treatment doses | Day 56
  Escalation in symptom control treatment doses will be defined as any escalation in the dose of a treatment existing at baseline or any new treatment introduced to control one of the following symptoms: pain, nausea, vomiting, lack of appetite, breathlessness, depression, anxiety, sleep disorders and wellness.
  The judgment criteria will be the proportion of patients with an escalation in symptom control treatment doses.
Number of side effects. | Day 7
  The number of side effects will be used to assess the security of use. It will be assessed using the Antidepressant Side Effect Checklist and side effects will be considered if rated moderate or severe.
Number of side effects. | Day 14
  The number of side effects will be used to assess the security of use. It will be assessed using the Antidepressant Side Effect Checklist and side effects will be considered if rated moderate or severe.
Number of side effects. | Day 28
  The number of side effects will be used to assess the security of use. It will be assessed using the Antidepressant Side Effect Checklist and side effects will be considered if rated moderate or severe.
Number of side effects. | Day 56
  The number of side effects will be used to assess the security of use. It will be assessed using the Antidepressant Side Effect Checklist and side effects will be considered if rated moderate or severe.
Medication adherence. | Day 56
  The medication adherence will be assessed using the Medication Adherence Rating Scale score at day 56 and the Proportion of Days Covered all along the follow-up period.
Symptoms' intensities auto-assessment on the following symptoms: pain, nausea, vomiting, lack of appetite, breathlessness, depression, anxiety, sleep disorders and wellness. | Day 28
  The Edmonton Symptom Assessment Scale 12F will be used to assess each symptoms intensities for the following symptoms: pain, nausea, vomiting, lack of appetite, breathlessness, depression, anxiety, sleep disorders and wellness.
  For each symptom, the difference between baseline and the assessment time will be used as the judgment criteria. A difference equal or over one point will be regarded as clinically significant.
Symptoms' intensities auto-assessment on the following symptoms: pain, nausea, vomiting, lack of appetite, breathlessness, depression, anxiety, sleep disorders and wellness. | Day 56
  The Edmonton Symptom Assessment Scale 12F will be used to assess each symptoms intensities for the following symptoms: pain, nausea, vomiting, lack of appetite, breathlessness, depression, anxiety, sleep disorders and wellness.
  For each symptom, the difference between baseline and the assessment time will be used as the judgment criteria. A difference equal or over one point will be regarded as clinically significant.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume ECONOMOS, MD, Principal Investigator — Centre Hospitalier Lyon Sud - Service de Soins Palliatifs
Locations (11):
- France (11):
  - Centre Hospitalier Universitaire de Clermont-Ferrand, Cébazat
  - Centre Hospitalier Universitaire de Grenoble, La Tronche
  - Hôpital Edouard Herriot, Lyon
  - Hôpital de la Croix-Rousse, Lyon
  - Centre Médico-Chirurgical de Réadaptation des Massues Croix-Rouge française, Lyon
  - Centre Léon Bérard, Lyon
  - Institut Curie, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Universitaire de Saint-Etienne, Saint-Etienne
  - Hôpitaux universitaires de Strasbourg, Strasbourg
  - Centre Hospitalier de Valence, Valence

REFERENCES:
- [Derived] Economos G, Alexandre M, Perceau-Chambard E, Villeneuve L, Subtil F, Haesebaert J, Glehen O. What is the effectiveness and safety of mirtazapine versus escitalopram in alleviating cancer-associated poly-symptomatology (the MIR-P study)? A mixed-method randomized controlled trial protocol. BMC Palliat Care. 2022 May 23;21(1):84. doi: 10.1186/s12904-022-00976-7. PMID 35599320